CLINICAL TRIAL: NCT04361188
Title: UPDRS-III Comparisons of Deep Brain Stimulation for Parkinson's Disease Between Patients Receiving MAC and AAA Anesthesia: a Randomized Controlled Trial
Brief Title: UPDRS-III Comparisons of DBS for PD Between Patients Receiving MAC and AAA Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, ZhiHeng Liu, Head of Anesthesiology, Shenzhen Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: FS20191119007
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease; Anesthesia
Keywords: Parkinson's disease; UPDRS-III; Deep Brain Stimulation; MAC; AAA
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAC anesthesia group (Experimental): Parkinson's disease patients receiving deep brain stimulation under MAC anesthesia.
  Interventions: Procedure: MAC anesthesia
- AAA anesthesia group (Active Comparator): Parkinson's disease patients receiving deep brain stimulation under AAA anesthesia.
  Interventions: Procedure: AAA anesthesia

INTERVENTIONS:
Procedure: MAC anesthesia — Patients receives DBS under monitored anesthesia care.
  Arms: MAC anesthesia group
Procedure: AAA anesthesia — Patients receives DBS under asleep-awake-asleep anesthesia.
  Arms: AAA anesthesia group

SUMMARY:
Compares the patients' scores of UPDRS-III before and six-month after receiving deep brain stimulation for Parkinson's disease under MAC or AAA anesthesia.

DETAILED DESCRIPTION:
Compares the patients' scores of UPDRS-III before and six-month after receiving deep brain stimulation for Parkinson's disease under MAC or AAA anesthesia. Besides, the research also compares the adverse events, LED, dosage of anesthetic drugs, wake-up time, surgical time, Hoehn&Yahr, PQD-39, MMSE, MoCA, HAMA, HAMD and patients' satisfaction between the two groups mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Diagnosis of primary Parkinson's disease
* Parkinson's disease-related symptoms remain difficult to control with appropriate anti-parkinsonian medications.

Exclusion Criteria:

* Refusal to Participate in the research
* Patients with severe comorbidities such as severe sleep apnea syndrome and metal disorder
* Previous functional neurosurgery: DBS, thalamic incision, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Scores' change of Unified Parkinson's Rating Scale (part III/motor part) | Before and six-month after DBS.
  Compares the scores' change of Unified Parkinson's Rating Scale (part III/motor part) between the two groups.

SECONDARY OUTCOMES:
Change of Levodopa Equivalent Dose | Before and six-month after DBS.
  Compares the change of Levodopa equivalent dose between the two groups.
Rates of Adverse Events | Intra-operative.
  Compares the rates of adverse events between the two groups.
Dosage of Anesthetic Drugs | Within surgery.
  Compares the dosage of anesthetic between the two groups.
Wake-up Time | Within surgery.
  Compares the wake-up time between the two groups.
Surgical Time | Within surgery.
  Compares the surgical time between the two groups.
Hoehn&Yahr | Before surgery.
  Compares the Hoehn&Yahr classification between the two groups' patients.
Patients' Satisfaction(Visual Analogue Scale) | 24 hours after surgery.
  Compares the scores of patients' satisfaction between the two groups' patients by Using a visual analogue scale. The minimum value is 0 and maximum value is 10. Higher value means greater satisfaction.
Scores' change of 39-item Parkinson's Disease Questionnaire | Before and six-month after DBS.
  Compares the scores' change of 39-item Parkinson's Disease Questionnaire between the two groups.
Scores' change of Mini-mental State Examination | Before and six-month after DBS.
  Compares the scores' change of Mini-mental State Examination between the two groups.
Scores' change of Montreal Cognitive Assessment | Before and six-month after DBS.
  Compares the scores' change of Montreal Cognitive Assessment between the two groups.
Scores' change of Hamilton Anxiety Scale | Before and six-month after DBS.
  Compares the scores' change of Hamilton Anxiety Scale between the two groups.
Scores' change of Hamilton Depression Scale | Before and six-month after DBS.
  Compares the scores' change of Hamilton Depression Scale between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhiheng, Doctor, Study Chair — Anesthesia department of Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ho AL, Pendharkar AV, Brewster R, Martinez DL, Jaffe RA, Xu LW, Miller KJ, Halpern CH. Frameless Robot-Assisted Deep Brain Stimulation Surgery: An Initial Experience. Oper Neurosurg. 2019 Oct 1;17(4):424-431. doi: 10.1093/ons/opy395. PMID 30629245
- [Result] Kulikov A, Lubnin A. Anesthesia for awake craniotomy. Curr Opin Anaesthesiol. 2018 Oct;31(5):506-510. doi: 10.1097/ACO.0000000000000625. PMID 29994938
- [Result] Krauss P, Marahori NA, Oertel MF, Barth F, Stieglitz LH. Better Hemodynamics and Less Antihypertensive Medication: Comparison of Scalp Block and Local Infiltration Anesthesia for Skull-Pin Placement in Awake Deep Brain Stimulation Surgery. World Neurosurg. 2018 Dec;120:e991-e999. doi: 10.1016/j.wneu.2018.08.210. Epub 2018 Sep 7. PMID 30196173
- [Result] Kochanski RB, Sani S. Awake versus Asleep Deep Brain Stimulation Surgery: Technical Considerations and Critical Review of the Literature. Brain Sci. 2018 Jan 19;8(1):17. doi: 10.3390/brainsci8010017. PMID 29351243
- [Result] Ho AL, Ali R, Connolly ID, Henderson JM, Dhall R, Stein SC, Halpern CH. Awake versus asleep deep brain stimulation for Parkinson's disease: a critical comparison and meta-analysis. J Neurol Neurosurg Psychiatry. 2018 Jul;89(7):687-691. doi: 10.1136/jnnp-2016-314500. Epub 2017 Mar 1. PMID 28250028
- [Result] Chen T, Mirzadeh Z, Chapple KM, Lambert M, Shill HA, Moguel-Cobos G, Troster AI, Dhall R, Ponce FA. Clinical outcomes following awake and asleep deep brain stimulation for Parkinson disease. J Neurosurg. 2018 Mar 16;130(1):109-120. doi: 10.3171/2017.8.JNS17883. Epub 2018 Mar 16. PMID 29547091
- [Result] Chen T, Mirzadeh Z, Chapple KM, Lambert M, Evidente VGH, Moguel-Cobos G, Oravivattanakul S, Mahant P, Ponce FA. Intraoperative test stimulation versus stereotactic accuracy as a surgical end point: a comparison of essential tremor outcomes after ventral intermediate nucleus deep brain stimulation. J Neurosurg. 2018 Aug;129(2):290-298. doi: 10.3171/2017.3.JNS162487. Epub 2017 Oct 13. PMID 29027853
- [Result] Sheshadri V, Rowland NC, Mehta J, Englesakis M, Manninen P, Venkatraghavan L. Comparison of General and Local Anesthesia for Deep Brain Stimulator Insertion: A Systematic Review. Can J Neurol Sci. 2017 Nov;44(6):697-704. doi: 10.1017/cjn.2017.224. Epub 2017 Sep 18. PMID 28920562
- [Result] Grant R, Gruenbaum SE, Gerrard J. Anaesthesia for deep brain stimulation: a review. Curr Opin Anaesthesiol. 2015 Oct;28(5):505-10. doi: 10.1097/ACO.0000000000000230. PMID 26308514
- [Result] Erickson KM, Cole DJ. Anesthetic considerations for awake craniotomy for epilepsy and functional neurosurgery. Anesthesiol Clin. 2012 Jun;30(2):241-68. doi: 10.1016/j.anclin.2012.05.002. Epub 2012 Jul 3. PMID 22901609
- [Result] Bronstein JM, Tagliati M, Alterman RL, Lozano AM, Volkmann J, Stefani A, Horak FB, Okun MS, Foote KD, Krack P, Pahwa R, Henderson JM, Hariz MI, Bakay RA, Rezai A, Marks WJ Jr, Moro E, Vitek JL, Weaver FM, Gross RE, DeLong MR. Deep brain stimulation for Parkinson disease: an expert consensus and review of key issues. Arch Neurol. 2011 Feb;68(2):165. doi: 10.1001/archneurol.2010.260. Epub 2010 Oct 11. PMID 20937936